CLINICAL TRIAL: NCT00173693
Title: What is the Best Policy to Prevent Osteoporotic Fracture?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9461700347
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-11

CONDITIONS: Osteoporosis or Osteopenia
Keywords: CEA, Osteoporosis, Fracture, Prevention, Exercise
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Fractures, Bone; Motor Activity | interventions — Exercise

INTERVENTIONS:
Behavioral: exercise for strength, balance, health education

SUMMARY:
This study aims to conduct a cost-effectiveness analysis (CEA) among the programs for preventing osteoporotic fracture. The main comparison will be made among the effects of three programs for preventing osteoporotic fractures: 1. health education; 2. exercise intervention for enhancing bone mineral density (BMD); 3. exercise intervention for preventing falls. The "cost" will be measured bases on the monetary cost of implementation of each program. The "effectiveness" will be measured includes the number of prevented osteoporotic fractures of each program, and related outcomes are the follows: 1. the medical cost of osteoporotic fracture; 2. the change of BMD in consecutive years; 3. the quality of life (QOL) of patients with osteoporotic fracture as compared to the reference population.

DETAILED DESCRIPTION:
This study aims to conduct a cost-effectiveness analysis (CEA) among the programs for preventing osteoporotic fracture. The main comparison will be made among the effects of three programs for preventing osteoporotic fractures: 1. health education; 2. exercise intervention for enhancing bone mineral density (BMD); 3. exercise intervention for preventing falls. The "cost" will be measured bases on the monetary cost of implementation of each program. The "effectiveness" will be measured includes the number of prevented osteoporotic fractures of each program, and related outcomes are the follows: 1. the medical cost of osteoporotic fracture; 2. the change of BMD in consecutive years; 3. the quality of life (QOL) of patients with osteoporotic fracture as compared to the reference population.

First year (2006): mainly a preparation stage

1. To conduct a meta-analysis of the effects of various interventions of prevention of osteoporotic fracture, especially in exercise models.
2. To establish the exercise programs for the intervention in the 2nd year, including the booklets and the posters.
3. To review the other alternatives of prevention of osteoporotic fracture.
4. To establish the social network needed for the following research. Second year (2007): to start the community-based field studies in Neihu District, Taipei.

All 37 "Lis" in Neihu will be invited to join the study, but only the Lis with willingness of participation will be the units for cluster sampling, and will be randomized to the three programs (Li as a unit). People living in the sampled Lis meet the inclusion criteria (postmenopausal (minimum for 1year) women and men over 65 years old) will be recruited and they will be further randomized into intervention group or reference group within each program.

1.To collect the baseline data. Baseline data include: the BMD, physical activity, nutrition diary, muscle strength, balance, risk factors of osteoporosis, history of fractures and falls 2.To execute the interventions. Three programs will be executed in the sampled Lis. They are all designed as a randomized control trial.

1. Health education (HE trial): lectures on knowledge of osteoporosis, osteoporotic fracture, the risk factors, the nutritional demand, the exercise principles for enhancing BMD and preventing fall.
2. Intervention for enhancing BMD (BMD trial): interventions to emphasize on weight-bearing exercise and trunk stabilization exercises. The exercise program will be supervised by a professional physical therapist 3 times per week for 3 months.
3. Intervention for preventing falls (fall prevention trial): interventions to emphasize on balance and strength training exercises. The exercise program will be also supervised by a professional physical therapist 3 times per week for 3 months.

   3.To apply the NHRI released health insurance data (2002-2006) for the next year study Third year (2008): follow-up, cost calculation and study on medical cost
   1. To calculate the cost of three intervention programs (from the view of provider).
   2. Telephone follow-up (FU) and recording the incidence of fall & fracture every 3 months.
   3. The first FU (1st FU) of the items collected at baseline.
   4. To study the medical cost of osteoporotic fracture with NHRI data. Fourth year (2009): continuing follow-up and study on QOL

   <!-- -->

   1. Continuing the telephone FU and recording the incidence of fall & fracture every 3 months
   2. The second FU (2nd FU) of the items collected at baseline
   3. To conduct a survey for the health-related QOL of people with osteoporotic fracture from outpatient clinics in hospital and the newly fractured subjects in the community.

   Fifth year (2010): continuing follow-up and CEA
   1. Continuing the telephone FU and recording the incidence of fall & fracture every 3 months.
   2. The third FU (3rd F/U) of the items collected at baseline.
   3. To investigate the effects of each intervention program

ELIGIBILITY:
Inclusion Criteria:

* post menopausal women or male over 65 y/o

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density, osteoporotic fracture

SECONDARY OUTCOMES:
CEA, Osteoporosis, Fracture, Prevention, Exercise

CONTACTS AND LOCATIONS:
Overall Officials: J Y Tsauo, PhD, Study Director — Grad School of PT, College of Medicine, NTU
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan